CLINICAL TRIAL: NCT06548984
Title: Respiratory Sarcopenia in Older Adults: Prevalence, Associated Factors and Response to an Exercise Program
Brief Title: Respiratory Sarcopenia in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Felipe León Morillas (Other)
Responsible Party: Sponsor-Investigator, Felipe León Morillas, Investigator, Catholic University of Murcia
Organization: Catholic University of Murcia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SarcoResp_Com
Record Dates: First submitted 2024-03-07; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Sarcopenia
Keywords: Sarcopsarcopenia; geriatrics; respiratory function
MeSH Terms: conditions — Sarcopenia; Respiratory Aspiration | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): diaphragmatic exercises
  Interventions: Other: diaphragmatic exercises
- Experimental group 2 (Experimental): Respiratory muscle training
  Interventions: Other: Respiratory muscle training
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: diaphragmatic exercises — Perform controlled and supervised diaphragmatic exercises
  Arms: Experimental group 1
Other: Respiratory muscle training — Perform respiratory muscle training with controlled and supervised devices
  Arms: Experimental group 2

SUMMARY:
The objectives of this study are to describe the prevalence of respiratory sarcopenia, evaluate its pattern of evolution over a one-year follow-up, and determine the response to a therapeutic exercise program in older adults in a geriatric nursing clinic.

A sample of approximately 115 older adults, of both sexes, from the geriatric nursing clinic of the Virgen de la Arrixaca Hospital, Murcia, will participate in the study. In the first stage, a prospective observational study will be carried out, with one year of follow-up, and subsequently a randomized controlled clinical trial, with patients who have been diagnosed with respiratory sarcopenia. In the clinical trial, patients will be divided into 3 groups: control, experimental 1 (diaphragmatic exercises) and experimental 2 (respiratory muscle training). Sociodemographic and clinical variables, physical function (palm grip, 5STS, 4MGS), respiratory function (respiratory muscle strength and diaphragmatic thickness) and health outcomes (respiratory infections, visit to the emergency department, hospitalization, falls, bedridden and/or death). Descriptive statistics, univariate and multivariate logistic regression models, Cox proportional hazards model and Kaplan-Meier curves will be used to analyze the data from the longitudinal study. To compare the differences between pre- and post-intervention of the clinical trial, a two-factor analysis of variance for repeated measures will be used. A P-value <0.05 will be considered significant in all analyses. The recording and analysis of the data will be carried out with the IBM SPSS Statistics 24® program.

ELIGIBILITY:
Inclusion Criteria:

* have functional ambulation (even with technical aids)
* be able to obey simple commands, such as taking deep breaths
* have sufficient oral occlusion capacity to perform respiratory tes

Exclusion Criteria:

* presence of acute respiratory diseases
* serious orthopedic diseases that interfere with measurements
* diagnosis of severe dementia
* those who present any contraindication for performing respiratory pressure measurement tests, as established in the guidelines of the Spanish Society of Pulmonology and Thoracic Surgery (SEPAR).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
RESPIRATORY MUSCLE FUNCTION | 24 Months
  INSPIRATORY AND EXPIRATORY PRESSURE OF THE MUSCULATURE
ultrasound | 24 Months
  diaphragm muscle thickness
physical function hand grip | 24 Months
  Hand grip: palm press strength
Physical function | 24 Months
  five times sit-up test (5STS)
Physical function walking speed | 24 Months
  walking speed (4MGS)
body composition | 24 Months
  Calculation of bioimpedance

SECONDARY OUTCOMES:
Sociodemografic | 24 months
  sex, age, marital status and educational level

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic Virgen de la Arrixaca Ctra. Madrid-Cartagena, s/n, 30120 El Palmar, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Background] Beaudart C, Zaaria M, Pasleau F, Reginster JY, Bruyere O. Health Outcomes of Sarcopenia: A Systematic Review and Meta-Analysis. PLoS One. 2017 Jan 17;12(1):e0169548. doi: 10.1371/journal.pone.0169548. eCollection 2017. PMID 28095426
- [Background] Papadopoulou SK, Tsintavis P, Potsaki P, Papandreou D. Differences in the Prevalence of Sarcopenia in Community-Dwelling, Nursing Home and Hospitalized Individuals. A Systematic Review and Meta-Analysis. J Nutr Health Aging. 2020;24(1):83-90. doi: 10.1007/s12603-019-1267-x. PMID 31886813
- [Background] Tovar-Alcaraz A, de Oliveira-Sousa SL, Leon-Garzon MC, Gonzalez-Carrillo MJ. [Effects of inspiratory muscle training on respiratory function and balance in stroke survivors: a randomized controlled trial]. Rev Neurol. 2021 Feb 16;72(4):112-120. doi: 10.33588/rn.7204.2020532. Spanish. PMID 33570158
- [Background] de Oliveira-Sousa SL, Leon-Garzon MC, Gacto-Sanchez M, Ibanez-Vera AJ, Espejo-Antunez L, Leon-Morillas F. Does Inspiratory Muscle Training Affect Static Balance in Soccer Players? A Pilot Randomized Controlled Clinical Trial. Healthcare (Basel). 2023 Jan 14;11(2):262. doi: 10.3390/healthcare11020262. PMID 36673630